CLINICAL TRIAL: NCT07248917
Title: A Comparative Evaluation of Sevoflurane Consumption and Anesthetic Depth During the Initial Phase of Minimal-Flow Versus Low-Flow Anesthesia in Patients Undergoing Retrograde Intrarenal Surgery (RIRS)
Brief Title: Evaluation of Sevoflurane Consumption During Initial Phase of Minimal-Flow Anesthesia in Retrograde Intrarenal Surgery
Acronym: SEVOMIN-RIRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Umit Yildiz, Medical Doctor in Anesthesiology and Reanimation, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KLKSH-ANES-SEVOMIN-RIRS-001; 2024/16/925 (Other: T.C. Sağlık Bilimleri Üniversitesi Kartal Dr. Lütfi Kırdar Eğitim ve Araştırma Hastanesi)
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Retrograde Intrarenal Surgery (RIRS); Urolithiasis; Minimal-flow Anesthesia; Sevoflurane; Anesthetic Consumption; Inhalational Anesthesia; Anesthesia Depth Monitoring
Keywords: minimal-flow anesthesia, low-flow anesthesia, sevoflurane, retrograde intrarenal surgery (RIRS), volatile consumption, environmental sustainability, MAC, BIS
MeSH Terms: conditions — Urolithiasis; Mycobacterium avium-intracellulare Infection

STUDY DESIGN:
Intervention Model Description: This was a prospective, two-arm, parallel-group study in which patients undergoing retrograde intrarenal surgery (RIRS) were randomly assigned to receive either minimal-flow (0.5 L/min) or low-flow (1.0 L/min) sevoflurane anesthesia. Participants were allocated to one group only and followed independently throughout the procedure. No crossover between groups occurred. The study aimed to compare anesthetic consumption, depth of anesthesia, and cardiorespiratory safety between the two anesthetic flow techniques.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimal-flow Sevoflurane Group (Experimental): Participants in this group received general anesthesia using sevoflurane with a fresh gas flow rate reduced to 0.5 L/min after the initial 10 minutes of induction. Anesthesia depth was monitored using BIS, and agent consumption and respiratory parameters were recorded throughout the retrograde intrarenal surgery (RIRS) procedure.
  Interventions: Drug: Sevoflurane Anesthesia with Minimal-flow
- Low-flow Sevoflurane Group (Active Comparator): Participants in this group received general anesthesia using sevoflurane with a consistent 1.0 L/min fresh gas flow during the maintenance phase. BIS monitoring, agent consumption, and respiratory parameters were recorded throughout the retrograde intrarenal surgery (RIRS).
  Interventions: Drug: Sevoflurane Anesthesia with Low-flow

INTERVENTIONS:
Drug: Sevoflurane Anesthesia with Minimal-flow — Patients received general anesthesia with sevoflurane. After induction, the fresh gas flow rate was reduced to 0.5 L/min during the maintenance phase of anesthesia for retrograde intrarenal surgery (RIRS). Agent consumption and anesthetic depth (via BIS and MAC) were monitored.
  Arms: Minimal-flow Sevoflurane Group
Drug: Sevoflurane Anesthesia with Low-flow — Patients received general anesthesia with sevoflurane. A fresh gas flow rate of 1.0 L/min was maintained during the maintenance phase of anesthesia for retrograde intrarenal surgery (RIRS). BIS, MAC, and respiratory parameters were recorded.
  Arms: Low-flow Sevoflurane Group

SUMMARY:
This study aimed to compare the effects of minimal-flow (0.5 L/min) and low-flow (1.0 L/min) sevoflurane anesthesia on agent consumption, anesthetic depth, and cardiorespiratory safety during retrograde intrarenal surgery (RIRS). A total of 62 adult patients undergoing elective RIRS were enrolled in this single-center interventional trial. Patients were divided into two groups based on the fresh gas flow rate used during the maintenance phase of anesthesia. The primary outcome was total sevoflurane consumption at the end of anesthesia. Secondary outcomes included time to reach 1 minimum alveolar concentration (MAC), vaporizer shut-off time, BIS values, MAC levels, and respiratory parameters. The study found that minimal-flow anesthesia was as effective and safe as low-flow anesthesia, with lower agent consumption and no adverse effects on hemodynamic or respiratory parameters. These findings support the use of minimal-flow anesthesia for improved cost-efficiency and environmental sustainability.

DETAILED DESCRIPTION:
This prospective, single-center, interventional study was designed to evaluate and compare the effects of minimal-flow and low-flow anesthesia on sevoflurane consumption, anesthetic depth, and respiratory parameters during retrograde intrarenal surgery (RIRS). After obtaining ethics committee approval (Decision No: 2024/16/925, Date: 17.09.2024), a total of 62 adult patients undergoing elective RIRS under general anesthesia were enrolled and divided into two groups based on the fresh gas flow rate used during the maintenance phase of anesthesia.

In Group 1 (Minimal-flow group), the fresh gas flow was reduced to 0.5 L/min after the initial 10 minutes of anesthesia. In Group 2 (Low-flow group), a 1.0 L/min flow rate was maintained. Both groups received the same induction and maintenance protocols with sevoflurane, and depth of anesthesia was monitored via BIS (Bispectral Index). Key variables measured included the total amount of sevoflurane consumed (mL), the time to reach 1 MAC, the vaporizer shut-off time, intraoperative BIS and MAC values, EtCO₂, and respiratory rate. Safety outcomes such as hemodynamic stability and desaturation were also recorded.

The primary outcome was total sevoflurane consumption. Secondary outcomes included anesthetic depth consistency (BIS/MAC), respiratory parameters, and time-based metrics. Statistical analysis revealed that minimal-flow anesthesia significantly reduced sevoflurane usage without compromising patient safety or anesthetic depth.

The results support the clinical use of minimal-flow anesthesia as a safe, cost-effective, and environmentally favorable alternative to low-flow techniques in selected urological procedures.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years

ASA (American Society of Anesthesiologists) Physical Status I or II

Scheduled to undergo elective retrograde intrarenal surgery (RIRS) under general anesthesia

Provided written informed consent

Able to cooperate with preoperative evaluation procedures

Exclusion Criteria:

* ASA Physical Status III or higher

History of respiratory disease (e.g., asthma, COPD, restrictive lung disease)

Known hepatic or renal dysfunction

Neurological or psychiatric disorders that may affect BIS monitoring or anesthetic response

Known allergy or hypersensitivity to sevoflurane or other volatile anesthetics

Pregnancy or breastfeeding

Obesity (BMI > 30 kg/m²)

Anticipated difficult airway or history of intubation complications

Participation in another clinical trial within the past 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Total Sevoflurane Consumption (mL) | End of surgery (approximately 60-90 minutes after anesthesia induction)
  Total volume of sevoflurane (in milliliters) used during the maintenance phase of general anesthesia, calculated automatically by the anesthesia machine and recorded at the end of surgery.

OTHER OUTCOMES:
Time to Reach 1 MAC (minutes) | Intraoperative (within first 10 minutes of anesthesia)
  Time in minutes from anesthesia induction to reaching 1 Minimum Alveolar Concentration (MAC) of sevoflurane, as recorded by the anesthesia machine.
Vaporizer Shut-off Time (minutes) | Intraoperative
  Time in minutes from the start of surgery to the moment the sevoflurane vaporizer was turned off.
End-Tidal CO₂ (EtCO₂) Levels (mmHg) | Throughout surgery
  Mean and peak end-tidal CO₂ levels measured intraoperatively at 10-minute intervals.
BIS Values During Maintenance (BIS Index Units) | Throughout surgery
  Bispectral Index values recorded at 10-minute intervals during the maintenance phase of anesthesia to assess anesthetic depth.
MAC Values During Maintenance (MAC Units) | Throughout surgery
  MAC values recorded during anesthesia maintenance to assess depth and consistency of volatile agent effect.
Respiratory Rate (breaths per minute) | Throughout surgery
  Intraoperative respiratory rates monitored and recorded to assess ventilatory response under different flow settings.
Oxygen Saturation (SpO₂, %) | Throughout surgery
  Minimum oxygen saturation values recorded intraoperatively to evaluate respiratory safety.

CONTACTS AND LOCATIONS:
Overall Officials: UMIT YILDIZ, M.D., Principal Investigator — Department of Anesthesiology and Reanimation, Kartal Dr. Lütfi Kırdar City Hospital, University of Health Sciences, Istanbul, Turkey
Locations (1):
- Kartal Dr. Lütfi Kırdar City Hospital, University of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Our study is:
  Single-center
  Non-commercial
  Conducted as part of a medical specialty thesis
  There is no stated plan to share anonymized individual-level data beyond what is reported in our thesis or publication